CLINICAL TRIAL: NCT06385964
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Dose of SHR-4597 Inhalation in Healthy Subjects and Asthmatic Patients
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SHR-4597 Inhalation in Healthy Subjects and Asthmatic Patients
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-4597-101
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Healthy Subjects; Asthmatic Patients

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-4597 (Experimental)
  Interventions: Drug: SHR-4597
- SHR-4597 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR-4597 — SHR-4597 by dry powder inhalation
  Arms: SHR-4597
Drug: Placebo — Placebo by dry powder inhalation
  Arms: SHR-4597 Placebo

SUMMARY:
The primary objective of this randomized, double-blind, single/multiple ascending dose, placebo-controlled Phase I clinical trial was to evaluate the safety and tolerability of SHR-4597 in healthy subjects and asthmatic patients. The study consists of two parts: Part 1 involves single ascending inhalation dose in healthy subjects; Part 2 involves multiple ascending inhalation dose in asthmatic patients, further divided into Part 2A: multiple ascending inhalation dose in mild to moderate asthmatic patients, and Part 2B: multiple ascending inhalation dose in moderate to severe asthmatic patients. Subsequent lung pharmacokinetic studies of SHR-4597 inhalation will be conducted based on patients' PKPD data.

ELIGIBILITY:
Inclusion Criteria:

-

Healthy subjects:

* Understand the specific procedures of the trial, voluntarily participate in this trial, and sign the informed consent form in writing.
* Aged between 18 and 55 years old (inclusive of boundary values).
* Male subjects with a weight of ≥ 50 kg and female subjects with a weight of ≥ 45 kg, with a body mass index (BMI) between 18 and 30 kg/m2 (inclusive of boundary values).
* Vital signs, physical examinations, laboratory tests, chest X-rays, etc., are either normal or clinically insignificant in abnormalities.
* Female subjects of reproductive potential or male subjects whose partners are of reproductive potential must agree, from the time of signing the informed consent form until 1 month after the last dose of study drug administration, to have no plans for pregnancy and voluntarily adopt effective contraception measures (including partners), while also avoiding sperm/egg donation (see Appendix 1 for details).
* During the study period, participants must be able to comply with all study regulations and procedures and be able to use the inhalation device used in this study correctly.

Asthma patients:

* Age ≥ 18 years and ≤ 75 years, gender not specified.
* Body Mass Index (BMI) during screening period ≥ 18 and ≤ 30 kg/m2.
* History records and objective evidence of asthma diagnosis meeting current guidelines in the 12 months prior to randomization.
* Not received any asthma treatment or only used short-acting bronchodilators (SABA) on an as-needed basis in the 4 weeks prior to randomization; or received maintenance therapy with medium to high daily doses of inhaled corticosteroids (ICS) and/or other asthma control medications for at least 3 months prior to randomization, and the dosage regimen and asthma condition remained stable in the 4 weeks prior to randomization.
* FEV1 ≥ 60% or ≥40% and < 80% of predicted value before inhalation bronchodilator use during screening and baseline.
* FeNO value ≥ 25 ppb during screening and baseline.
* Female subjects of reproductive potential or male subjects whose partners are of reproductive potential must agree, from the time of signing the informed consent form until 1 month after the last dose of study drug administration, to have no plans for pregnancy and voluntarily adopt effective contraception measures (including partners), while also avoiding sperm/egg donation (see Appendix 1 for details).
* Voluntarily sign the informed consent form to participate in this study.

Exclusion Criteria:

-

Healthy subjects:

* Suffering from any clinically serious disease such as circulatory, endocrine, nervous, digestive, respiratory, hematological, immunological, psychiatric and metabolic abnormalities, or any other disease that might interfere with the study results;
* Previous history of malignant tumor;
* Current or recent (within 3 months) respiratory disease or a history of severe respiratory disease, and researchers assess that it may affect drug absorption or pose a safety risk;
* Patients with severe infection, severe trauma or major surgical operation within 3 months before administration; Patients who plan to undergo surgery during the trial period and within two weeks of its end;
* 12-lead ECG abnormalities are clinically significant or ECG QT interval (QTc) > 450 ms in male subjects and ECG QTc > 470 ms in female subjects;
* Screening for infectious diseases during the screening period, including positive results for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody, human immunodeficiency virus antibody, and syphilis treponema antibody;
* People with a suspected history of allergy to the investigational drug or any of the ingredients in the investigational drug, allergies or a history of severe drug allergy;
* Previous blood collection difficulties or can not tolerate venipuncture, such as fainting needle, fainting blood
* Had taken any prescription, over-the-counter, or Chinese herbal medicine within 14 days prior to taking the study drug, or within 5 half-lives of the drug at the time of screening; Plan to take non-study medications during the trial period.;
* Participants who have participated in clinical trials of any drug or medical device within 3 months prior to screening, or those still within 5 half-lives of a drug prior to screening (whichever is longer);
* Blood donation or blood loss ≥ 200 mL within 1 month prior to administration, or blood donation or blood loss ≥ 400 mL within 3 months prior to administration, or received blood transfusion within 8 weeks;
* Average smoking ≥ 5 cigarettes per day in the three months prior to administration; More than 15 g of alcohol per day on average in the month prior to administration (15 g of alcohol is equivalent to 450 mL of beer or 150 mL of wine or 50 mL of low-alcohol liquor);
* People who do not refrain from smoking, drinking or consuming caffeinated food or beverages (more than 8 cups, 1 cup = 250 mL) 2 days before administration and during the trial period; Those who cannot prohibit the consumption of grapefruit or grapefruit juice; And those who have special requirements for diet and cannot comply with a unified diet;
* Subjects who are pregnant (tested positive during screening or baseline pregnancy test) or who plan to become pregnant while breastfeeding or during the study;
* Participants with positive drug screening or alcohol breath test during screening visit/baseline visit;
* Other conditions deemed by the investigator as unsuitable for participation in this trial;

Asthma patients:

* Combined with clinically significant lung diseases, including but not limited to active pulmonary tuberculosis, bronchiectasis, atelectasis, idiopathic pulmonary fibrosis, bronchopulmonary aspergillosis, and chronic obstructive pulmonary disease (COPD);
* Malignant tumors diagnosed within 5 years prior to randomization (Excluding malignancies with low risk of metastasis and death, such as adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix);
* Combined with poorly controlled hypertension (systolic blood pressure ≥180mmHg, and/or diastolic blood pressure ≥110mmHg during screening) or uncontrolled severe cardiovascular and cerebrovascular disease;
* Known immunodeficiency;
* A history of infections requiring clinical intervention within 4 weeks prior to randomization, including but not limited to respiratory infections:
* Known parasitic infection within 6 months prior to randomization;
* Receiving a non-selective beta-blocker (e.g., propranolol) within 1 week prior to randomization;
* Blood donation or significant blood loss (≥400ml), or transfusion of blood products or immunoglobulin within 4 weeks prior to randomization;
* Received attenuated live vaccines within 4 weeks prior to randomization;
* Allergen immunotherapy was administered 8 weeks before randomization
* Used systemic immunosuppressive agents (including systemic corticosteroids for asthma treatment, and other systemic corticosteroids <3 days for conditions other than asthma), or immunomodulators, or biologics or Th2 cell cytokine inhibitors within 12 weeks prior to randomization or within 5 half-lives of the drug (whichever is longer, with reference to the drug's prescribing information; for drugs with unknown half-life, the 12 weeks prior to randomization is considered;
* Bronchial thermoplasty was performed within 1 year prior to randomization
* Planned surgical procedures during the study period, or other therapeutic measures deemed by the investigator to potentially affect the assessment of the subjects;
* The screening period or baseline laboratory tests showed significant abnormalities
* Prolonged ECG QTc interval (men >450ms, women >470ms) or other clinically significant abnormal results that may pose a significant safety risk to subjects during the screening period
* Screening period is still smoking or quit smoking less than 6 months, or previous smoking ≥10 pack years (pack years = number of years of smoking × number of packs per day)
* A history of drug use, alcohol abuse (average consumption of ≥14 units of alcohol per week: 1 unit = 285 mL for beer, or 25 mL for spirits, or 100 ml for wine) or drug abuse within 1 year prior to screening
* Participated in another clinical study and used investigational drugs containing active ingredients within 30 days prior to screening, or still within 5 half-lives of the investigational drug at the time of screening (whichever is longer).
* Subjects who are pregnant (screening or baseline blood pregnancy test positive) or who plan to become pregnant while breastfeeding or during the study
* People who are allergic to the drug or its excipients, allergic or have a history of severe drug allergy
* Other reasons deemed by the investigator as unsuitable for participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of inhalant adverse events after 4 days of single inhalation of SHR4597 in healthy subjects | 4 days for healthy subjects
Incidence and severity of inhalant adverse events after 16 days of multiple inhalation of SHR4597 in asthmatic patients, | 16 days for asthmatic patients.

IPD SHARING:
Plan to Share IPD: Undecided